CLINICAL TRIAL: NCT06138600
Title: Acceptability and Feasibility of Injectable Cabotegravir Pre-exposure Prophylaxis (PrEP) Versus Oral PrEP in Routine Care up to 15 Months in Private Pharmacies in South Africa
Acronym: AXIS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Professor Francois Venter, Executive Director: Ezintsha, University of Witwatersrand, South Africa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EZ-FV-035
Record Dates: First submitted 2023-10-17; First posted 2023-11-18 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections
Keywords: Pre-Exposure Prophylaxis (PrEP); Long Acting Injectable; Cabotegravir
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Tenofovir; Emtricitabine; Lamivudine

STUDY DESIGN:
Intervention Model Description: Adult (≥18 and ≤ 35 years old) male or female willing to access PrEP at the same pharmacy for up to 2 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cabotegravir Long Acting Injectable (Active Comparator): Investigational Product: Cabotegravir Dosage Formulation: 600 mg suspension for injection Route of Administration: Intra-muscular injection Dosing Instructions: 1 vial (600 mg) injected monthly for the initial visit (Month 1 and 2), then every 2 months thereafter (from Month 2 onwards)
  Interventions: Drug: Cabotegravir Injection [Apretude]
- Tenofovir disoproxil fumarate + Emtricitabine/Lamivudine (TDF/FTC[3TC]) (Active Comparator): Investigational Product: Tenofovir disoproxil fumarate / emtricitabine (or lamivudine) Dosage Formulation: 300 mg / 200 mg (300mg) fixed dose combination tablet Route of Administration: Oral Dosing Instructions: 1 tablet (300/200/ TDF/FTC) daily or (300/300/TDF/3TC) daily
  Interventions: Drug: Tenofovir disoproxil fumarate / emtricitabine (or lamivudine)

INTERVENTIONS:
Drug: Cabotegravir Injection [Apretude] — White to slightly pink free flowing suspension suspension for injection contained in a brown coloured vial. Each vial is for single use and does not require dilution prior to administration.
  Other Names: Apretude
  Arms: Cabotegravir Long Acting Injectable
Drug: Tenofovir disoproxil fumarate / emtricitabine (or lamivudine) — TDF/FTC is currently available as standard of care for PrEP in the public sector as per the department of health guidelines.
  Other Names: Tenemine
  Arms: Tenofovir disoproxil fumarate + Emtricitabine/Lamivudine (TDF/FTC[3TC])

SUMMARY:
This is a mixed methods study employing a convergence model triangulation design. Participants in the study will be sexually active young adults starting Pre-exposure Prophylaxis at private pharmacies, who will be offered either Cabotegravir Long-Acting Injectable, oral Pre-exposure Prophylaxis (TDF/FTC[3TC]), or Pre-exposure Prophylaxis deferment at each of their regular visits, with the option to switch between options for up to 15 months, with a final exit interview following the transition to standard-of-care. The number of study visits will vary, depending on participant Pre-exposure Prophylaxis choices. Those choosing oral Pre-exposure Prophylaxis will be seen 3 monthly from V2 onwards, but those choosing Cabotegravir Long-Acting Injectable will be seen 2 monthly from V2. A maximum of 9 visits is possible.

DETAILED DESCRIPTION:
In the ATLAS study participants were asked, after they had transitioned back to conventional oral antiretroviral therapy, whether they preferred injectable or oral treatment. Their feedback on their preference overwhelming favoured injectables9. Women and men will be recruited from existing Ezintsha programs operating within the pharmacies, using current government criteria for Pre-exposure Prophylaxis initiation. Pre-exposure Prophylaxis will be initiated and monitored according to these and the Pharmacist-Initiated Management of Antiretroviral Therapy guidelines. Pre-exposure Prophylaxis, through these programs, will be offered free of charge. The study is designed to be as "real-world" as possible. Adaptations to routine Pre-exposure Prophylaxis guidelines have been made to accommodate visit-based HIV testing (based on the injectable regimens, which require more frequent access to the clinic). Participant reimbursement will therefore be for the baseline, mid and end-of-study interviews in participants consenting to these interviews. The maximum amount of time a participant in the study can be on either Cabotegravir Long-Acting Injectable or oral Pre-exposure Prophylaxis, or a combination, or, indeed, on neither drug, is therefore 15 months (and an additional three months on oral Pre-exposure Prophylaxis during the transition, as standard of care).

The Investigator anticipates that participants will favour Cabotegravir Long-Acting Injectable, but also anticipates that there may be interesting patterns of use when they learn that they may defer access to Cabotegravir Long-Acting Injectable or oral Pre-exposure Prophylaxis. Participants may favour Pre-exposure Prophylaxis, as they may prefer three monthly visits over the two monthly injection requirements. The Investigator may see participants initially choosing oral Pre-exposure Prophylaxis, and then moving to Cabotegravir Long-Acting Injectable, or even vice versa. The Investigator is unclear on what men may favour versus women. The Investigator will endeavor to recruit at least 20 men in the study, appreciating that not much is known about this group in the sub-Saharan Africa context. One of the most important analyses that will flow from information collected when assessing for Pre-exposure Prophylaxis eligibility is the risk profile of the participants taking up Pre-exposure Prophylaxis, a key issue when assessing cost-effectiveness. Finally, the investigator is not excluding women or men who defer Pre-exposure Prophylaxis initially. These various combinations will provide interesting quantitative, but more importantly, qualitative data on preferences, and on how services may be improved to accommodate participants' choices.

ELIGIBILITY:
Inclusion Criteria:

-

Each participant must meet all of the following criteria to be enrolled in this study:

1. Adult male or female (≥18 and ≤ 35 years old)
2. Is self-reported sexually active
3. HIV negative at the time of study enrolment (as determined by a rapid blood test for HIV 1)
4. Body weight ≥ 35 kilograms.
5. Creatinine clearance ≥ 60 mL/min.
6. Willingness to sign informed consent.

Exclusion Criteria:

-

Participants meeting the following criteria will be excluded from participating in the study:

1. Symptoms of HIV seroconversion (see Table 1).
2. Pregnant (participant must have a negative beta human chorionic gonadotrophin (b-hCG) urine test at screening) or lactating women, or women intending to become pregnant or breastfeed during the study.
3. Is in good health, with no surgical or medical condition which may significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the volunteer or the objectives of the study or impair their ability to comply with the dosing schedule and/or protocol evaluations. The Investigator should make this determination in consideration of the volunteer's medical history. This including, but not limited to, the following: a. History of severe hepatic impairment, history of liver cirrhosis with or without viral hepatitis co-infection.

   b. Unstable or poorly controlled seizure disorder. c. History of coagulopathies, or current or anticipated need for chronic anticoagulation.

   d. Presence of a tattoo or other dermatological condition overlying the gluteus region which would realistically obstruct administration of an intramuscular injection.
4. Known hypersensitivity to or specific contraindications to the use of TDF or FTC/3TC or CABLA.
5. Hep B surface antigen positive or known active Hep B infection.
6. Is receiving or has received the following agents within 28 days prior to screening, and cannot discontinue their use for the duration of the study:

   1. tuberculosis therapy (i.e., rifampicin, rifapentine, rifabutin)
   2. anticoagulation agents;
   3. anti-convulsants (e.g. carbamazepine, oxcarbazepine, phenobarbital, phenytoin);
   4. herbal products (e.g. St John's Wort).
7. Concurrent use of PrEP from a different medical provider, other than the study site
8. Participant is judged by the Investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results.
9. Inability or unwillingness to be followed up for the study period, including plans to move out the study geographical area in the next 12 months or otherwise unable to participate in the study visits as determined by the PI.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
To describe acceptability of CAB-LA (Long-Acting Cabotegravir) PrEP, amongst different PrEP modalities, including PrEP deferment, in eligible men and women. | 15 Months
  Acceptability of CAB-LA (Long-Acting Cabotegravir) as determined by qualitative and quantitative assessment using piloted and validated semi-structured questionnaires for acceptability. (Quantitative data will be expressed as ratios)
To describe acceptability of CAB-LA (Long-Acting Cabotegravir) PrEP, amongst different PrEP modalities, including PrEP deferment, in eligible men and women. | 12 Months
  Acceptability of Intervention Measure (AIM)/ Intervention Appropriateness Measure/ (IAM), at 12 months and end of study. (Expressed as ratios where applicable)

SECONDARY OUTCOMES:
To describe feasibility of CAB-LA (Long-Acting Cabotegravir) PrEP implementation, amongst different PrEP modalities, including PrEP deferment, in eligible men and women. | 15 Months
  Feasibility of CAB-LA (Long-Acting Cabotegravir) as determined by qualitative and quantitative assessment using piloted or validated semi-structured questionnaires and on feasibility conducted with participants and healthcare workers.
To describe feasibility of CAB-LA (Long-Acting Cabotegravir) PrEP implementation, amongst different PrEP modalities, including PrEP deferment, in eligible men and women. | 12 Months
  Feasibility of Intervention Measure (FIM) completed by healthcare workers at exit and participants at 12 months and end of study.
To describe the association of socio-demographic factors, reported sexual behaviour, PrEP knowledge and previous PrEP use on PrEP choice. | 15 Months
  Tests of association between PrEP choice and selected predictor variables.
To describe the association of socio-demographic factors, reported sexual behaviour, PrEP knowledge and previous PrEP use on PrEP choice. | 12 Months
  Proportion of individuals who are using each type of PrEP collected at study start, month 12 and end of study.
To describe the uptake, persistence and patterns of transition on each form of PrEP. | 15 Months
  Attending all study visits/retention extracted from participant EDC (Electronic Data Capture) visit forms.
To describe a risk profile of those taking up both PrEP regimens, as well as those deferring PrEP. | 15 Months
  Willingness to take CAB-LA (Long-Acting Cabotegravir) for the entire study duration extracted from participant EDC forms
To describe a risk profile of those taking up both PrEP regimens, as well as those deferring PrEP. | 15 Months
  Willingness to take CAB-LA post study stop collected at end of study using semi-structured interviews.
To describe operational suggestions from the participants regarding how health services could be improved regarding better/more comfortable/faster/cheaper/other add-on sexual reproductive services. | 15 Months
  Extent to which the study staff could easily administer CAB-LA (Long-Acting Cabotegravir).
To describe the provider experiences and perceptions of CAB-LA (Long-Acting Cabotegravir) PrEP implementation, amongst different PrEP modalities, including PrEP deferment, in eligible men and women. | 15 Months
  Healthcare worker perspectives on maintenance, demand creation and service delivery post study completion collected during a focus group discussion conducted at the end of the study.
To describe participant willingness-to-pay for PrEP services at the end of the study. | 15 Months
  Willingness to pay for CAB-LA (Long-Acting Cabotegravir) collected at the end of the study using semi-structured interviews.

OTHER OUTCOMES:
To describe patient reported and clinical significant adverse events of CAB LA (Long-Acting Cabotegravir) and oral PrEP(TDF/FTC[3TC]) over 15 months | 15 Months
  Reported incidence of SAEs (Serious Adverse Events) and DAIDS-defined Grade 3 and Grade 4 AEs, throughout study duration, including AEs considered related to the IMP and reported injection site reactions.
To describe patient reported and clinical significant adverse events of CAB LA (Long-Acting Cabotegravir) and oral PrEP(TDF/FTC[3TC]) over 15 months | 15 Months
  Proportion of participants reporting discontinuing treatment due to AEs (Adverse Events.
To describe patient reported and clinical significant adverse events of CAB LA (Long-Acting Cabotegravir) and oral PrEP(TDF/FTC[3TC]) over 15 months | 15 Months
  Proportion of participants scoring > 4 on AIM and IAM.
Viral integrase inhibitor resistance mutations in participants who seroconvert while on CAB-LA (Long-Acting Cabotegravir) PrEP will be documented. | 15 Months
  % of participants who seroconvert.
Viral integrase inhibitor resistance mutations in participants who seroconvert while on CAB-LA (Long-Acting Cabotegravir) PrEP will be documented. | 15 Months
  ART (Antiretroviral) resistance genotyping done if seroconversion occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Francois WD Venter, MBBCh, Study Director — Ezintsha, a division of Wits Health Consortium; Simiso M Sokhela, MBBCh, Principal Investigator — Ezintsha, a division of Wits Health Consortium; Nonkululeko M Mashabane, BPharm, Study Chair — Ezintsha, a division of Wits Health Consortium
Locations (1):
- Ezintsha, a division of Wits Health Consortium, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared is all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication
Access Criteria: Anyone who wishes to access the data